CLINICAL TRIAL: NCT03111160
Title: Lower Femtosecond Laser Energy Levels Lead to Better Visual Recovery After Small-incision Lenticule Extraction for Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-0840
Record Dates: First submitted 2017-03-26; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Myopia
Keywords: Small-incision lenticule extraction; femtosecond laser; lower laser energy level; early visual recovery
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Based on the review of literature, we regarded SMILE using energy levels of 115 nJ or higher as 'conventional' energy-SMILE (C-SMILE). Since 500kHz VisuMax femtosecond laser used in this study had a threshold photodisruption energy level of 100 nJ, lowest energy level of L-SMILE was set at 100 nJ. Because the spot distance must be changed by approximately 1 μm when laser energy changed by 50 nJ, we could set the maximum laser energy to 150 (100 + 50) nJ as highest one of C-SMILE while keeping the spot distance constant. Finally, we established two groups divided by different laser energies: L-SMILE group using lower energy levels of 100, 105, and 110 nJ, and C-SMILE group using 'conventional', not higher, energy levels of 115 to 150 nJ.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lower energy (Experimental): SMILE procedure using lower energy (100, 105, and 110 nJ)
  Interventions: Procedure: SMILE procedure using lower energy (100, 105, and 110 nJ)
- conventional energy (115 to 150 nJ) (Active Comparator): SMILE procedure using conventional energy (115 to 150 nJ)
  Interventions: Procedure: SMILE procedure using conventional energy (115 to 150 nJ)

INTERVENTIONS:
Procedure: SMILE procedure using lower energy (100, 105, and 110 nJ) — Based on the review of literature, we regarded SMILE using energy levels of 115 nJ or higher as 'conventional' energy-SMILE (C-SMILE). Since 500kHz VisuMax femtosecond laser used in this study had a threshold photodisruption energy level of 100 nJ, lowest energy level of L-SMILE was set at 100 nJ. Because the spot distance must be changed by approximately 1 μm when laser energy changed by 50 nJ, we could set the maximum laser energy to 150 (100 + 50) nJ as highest one of C-SMILE while keeping the spot distance constant. Finally, we established two groups divided by different laser energies: L-SMILE group using lower energy levels of 100, 105, and 110 nJ, and C-SMILE group using 'conventional', not higher, energy levels of 115 to 150 nJ.
  Arms: lower energy
Procedure: SMILE procedure using conventional energy (115 to 150 nJ) — The SMILE procedures were conducted in the Eyereum Eye Clinic (Seoul, South Korea). The target postoperative refraction was emmetropia. The surgery, using standardized techniques, was performed by an experienced surgeon (D.S.Y.K.) using the VisuMax system. The surgical parameters used during SMILE were as follows: repetition rate of 500 kHz, pulse energy 100 to 150 nJ (100, 105, and 110 nJ, L-SMILE; 115 to 150 nJ, C-SMILE), spot distance 4.5 μm (regardless of FSL energy), cap thickness 120 μm, and side-cut width 2 mm in the 12-o'clock position with an angle of 90°. After the anterior (upper) and posterior (lower) delineated plane of the intrastromal lenticule were well defined, the anterior and posterior interface were dissected with a micro-spatula with a blunt circular tip and extracted with micro-forceps. The integrity of the lenticule was also checked subsequently.
  Arms: conventional energy (115 to 150 nJ)

SUMMARY:
Small-incision lenticule extraction (SMILE), the most recently developed refractive surgical technique, is being performed in a growing number of cases. This intrastromal keratomileusis using only a femtosecond laser is a new procedure that extracts the refractive lenticule through a small corneal incision ranging from 2 to 5 mm, with the absence of a flap and the preservation of the anterior-most stromal lamellae and Bowman's layer (except for the region of the small incision). Many studies have demonstrated that SMILE achieved comparable or superior efficacy, safety, and predictability to femtosecond laser -assisted in situ keratomileusis (FS-LASIK) and femtosecond lenticule extraction (FLEx). However, the recovery of visual acuity in the early postoperative period after SMILE is slower, compared to other refractive surgery techniques. Therefore, adjusting energy might improve postoperative visual acuity and recovery time after SMILE. Nevertheless, the optimal parameters drawn from a well-organized randomized study have yet to be elucidated. The purpose of this study was to investigate the optimal femtosecond laser energy, with the aim of improving clinical outcomes during the early postoperative period after SMILE for the correction of myopia. To this end, we used a 500 kHz VisuMax with spot-spacing control at energy levels lower than 115 nJ, based on the previous studies. Therefore, we prospectively compared visual outcomes of two groups randomly divided by different laser energies: one underwent SMILE using lower energy levels of 100, 105, and 110 nJ (L-SMILE), while the other group underwent SMILE at energy levels conventionally used of 115 to 150 nJ (C-SMILE).

DETAILED DESCRIPTION:
This prospective randomized comparative study was approved by the Institutional Review Board, Yonsei University College of Medicine, Seoul, South Korea (IRB No. 4-2016-0840). The study adhered to the tenets of the Declaration of Helsinki and followed good clinical practices. All patients provided informed consent after a detailed explanation of the possible risks and benefits of the study. The right eye of each patient was included in the study unless contraindicated, in which case the left eye was used. The patients were randomized to one of two groups (L-SMILE or C-SMILE) by means of permuted block-randomization with the Clinstat software (Available from: http://www-users.york.ac.uk/~mb55/soft/soft.htm). Thereafter, the patients were randomly allocated a laser energy level within their SMILE group by means of minimization with the Minim software (Available from: http://www.users.york.ac.uk/~mb55/guide/minim.htm) due to the small sample size (< 200).

Patients were recruited from November 2016 to December 2017. All patients underwent a baseline preoperative assessment including anterior and posterior segment examinations. Inclusion criteria were: corneal thickness of more than 500 μm, manifest refractive sphere of -3.00 to -6.00 diopters (D), manifest refractive cylinder less than 6.00 D, stable refractive error with less than a 0.50 D change in sphere and cylinder in the previous year, corrected distance visual acuity (CDVA) of 20/20 or better in both eyes, and age of 20 years or older. Exclusion criteria were: severe ocular surface disease, any corneal disease, cataract, glaucoma, macular disease, or previous history of intraocular or corneal surgery. Patients with suspicion of keratoconus on corneal topography were also excluded.

We reviewed thoroughly literatures which included 239 online-available papers about SMILE, and, of them, we selected 116 original articles on clinical outcome or studies involving human lenticules after SMILE surgery and identified all the energy levels used in each article, as possible. Finally, we found almost all previous researches provided surgical results by using a 200 or 500 kHz VisuMax (Carl Zeiss Meditec AG, Jena, Germany) with energy levels of 115 to 190 nJ except only three studies: two studies by same researchers obscured the laser energy level (approximately 110 nJ) used in SMILE, however the other latest study provided definitely their laser energy 100 nJ (Figure 1 and supplemental table 1). There were 5 studies on SMILE using 115 nJ of laser energy in the literature.

Based on the review of literature, we regarded SMILE using energy levels of 115 nJ or higher as 'conventional' energy-SMILE (C-SMILE). Since 500kHz VisuMax femtosecond laser used in this study had a threshold photodisruption energy level of 100 nJ, lowest energy level of L-SMILE was set at 100 nJ. Because the spot distance must be changed by approximately 1 μm when laser energy changed by 50 nJ, we could set the maximum laser energy to 150 (100 + 50) nJ as highest one of C-SMILE while keeping the spot distance constant. Finally, we established two groups divided by different laser energies: L-SMILE group using lower energy levels of 100, 105, and 110 nJ, and C-SMILE group using 'conventional', not higher, energy levels of 115 to 150 nJ.

Based on our preliminary results (n=6 per group) showing the significant mean difference of postoperative visual acuity between C-SMILE and L-SMILE, a priori power analysis was performed. Group sample sizes of 54 and 81 achieved 81% power to detect a difference of - 0.1 between the null hypothesis that both group means are 0.0 and the alternative hypothesis that the mean of group 2 is 0.1 with estimated group standard deviations of 0.1 and 0.1 and with a significance level (alpha) of 0.05 using a two-sided two-sample t-test. Therefore, we confirmed that sample size of L-SMILE is 60 and one of C-SMILE is 90 as considering 10 % reduction.

ELIGIBILITY:
Inclusion Criteria:

1. age of 20 years or older.
2. corneal thickness of more than 500 μm
3. manifest refractive sphere of -3.00 to -6.00 diopters (D)
4. manifest refractive cylinder less than 6.00 D
5. stable refractive error with less than a 0.50 D change in sphere and cylinder in the previous year
6. corrected distance visual acuity (CDVA) of 20/20 or better in both eyes

Exclusion Criteria:

1. severe ocular surface disease
2. any corneal disease, cataract, glaucoma, macular disease, or previous history of intraocular or corneal surgery
3. Patients with suspicion of keratoconus on corneal topography

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Uncorrected Distance Vision Acuity | within the first 90 days after surgery
  Uncorrected Distance Vision Acuity bya Snellen visual acuity chart
Corneal aberration | within the first 90 days after surgery
  Corneal aberration automatically recoreded by a wavefront analysis machine

SECONDARY OUTCOMES:
surface roughness of lenticules | immediately after SMILE surgery
  By atomic force microscopy, the average roughness (Ra, µm), root-mean-square roughness (Rq, µm), and ten-point mean height roughness (Rz, µm) are automatically recorded on the height images.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Yonsei Univeristy College of Medicine, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reinstein DZ, Archer TJ, Gobbe M. Small incision lenticule extraction (SMILE) history, fundamentals of a new refractive surgery technique and clinical outcomes. Eye Vis (Lond). 2014 Oct 16;1:3. doi: 10.1186/s40662-014-0003-1. eCollection 2014. PMID 26605350
- [Background] Wang JS, Xie HT, Jia Y, Zhang MC. Small-incision lenticule extraction versus femtosecond lenticule extraction for myopic: a systematic review and Meta-analysis. Int J Ophthalmol. 2017 Jan 18;10(1):115-121. doi: 10.18240/ijo.2017.01.19. eCollection 2017. PMID 28149787
- [Background] Donate D, Thaeron R. Lower Energy Levels Improve Visual Recovery in Small Incision Lenticule Extraction (SMILE). J Refract Surg. 2016 Aug 1;32(9):636-42. doi: 10.3928/1081597X-20160602-01. PMID 27598734